CLINICAL TRIAL: NCT04214626
Title: A Single-arm, Multi-center, Phase II Clinical Trial of R-CHOP Combined With Lenalidomide in the First-line Treatment for Patients With Medium to High Risk/High Risk Diffuse Large B Cell Lymphoma
Brief Title: R-CHOP Combined With Lenalidomide in the First-line Treatment for Patients With Diffuse Large B Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yanyan Liu, Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HNSZLYYNHL02
Record Dates: First submitted 2019-12-26; First posted 2020-01-02 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-04

CONDITIONS: Diffuse Large B Cell Lymphoma
Keywords: Diffuse Large B Cell Lymphoma; R-CHOP; Lenalidomide
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Rituximab; Lenalidomide; Cyclophosphamide; Epirubicin; Vincristine; Prednisone; Methotrexate

STUDY DESIGN:
Intervention Model Description: R-CHOP combined with Lenalidomide in the first-line treatment for patients with medium to high risk/high risk DLBCL.
  The individuals with the same propensity score according to high-risk factors (IPI score, double-expressor and P53 protein positive) were set as external control group (1:1) treated with R-CHOP.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- R-CHOP regimen Combined With Lenalidomide (Experimental): Experimental: R-CHOP regimen Combined With Lenalidomide Induction Chemotherapy: Rituximab, 375mg/m2, Intravenous administration on day 0, Lenalidomide, 25mg oral administration on day 1 to 10, combined with regimen：CHOP (Cyclophosphamide, Epirubicin, Vincristine and Prednisone): repeated every 3 weeks, up to 6 cycles.
  Patients will exit and receive salvage treatment for the following situations: disease progression, stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops.
  Maintenance Treatment for patients with CR after 6 cycles: Rituximab, 375mg/m2, Intravenous administration on day 0 repeated every 3 weeks until disease progression or unacceptable toxicity develops, up to 2 cycles.
  PS: Methotrexate, 1g/m2, Intravenous administration on day 3 of each 3-week cycle, from 2 to 5 cycles for patients with high recurrence risk of the central nervous system.
  Interventions: Drug: Rituximab; Drug: Lenalidomide; Drug: Cyclophosphamide; Drug: Epirubicin; Drug: Vincristine; Drug: Prednisone; Drug: Methotrexate

INTERVENTIONS:
Drug: Rituximab — Induction Chemotherapy: 375mg/m2, Intravenous administration on day 0 of each 3-week cycle until disease progression, stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Maintenance Treatment for patients with CR after 6 cycles: Rituximab, 375mg/m2, Intravenous administration on day 0 repeated every 3 weeks until disease progression or unacceptable toxicity develops, up to 2 cycles (Total 8 cycles).
  Other Names: RiTUXimab Injection
Drug: Lenalidomide — Induction Chemotherapy: 25mg, oral administration on day 1 to 10 of each 3-week cycle until disease progression, stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Lenalidomide capsule
Drug: Cyclophosphamide — Induction Chemotherapy: 750mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression, stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Cyclophosphamide Injection
Drug: Epirubicin — Induction Chemotherapy: 70mg/m2, Intravenous administration on day 1 of each 3-week cycle until disease progression, stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Epirubicin hydrochloride
Drug: Vincristine — Induction Chemotherapy: 1.4mg/m2 (Max: 2mg), Intravenous administration on day 1 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Vincristine Injection
Drug: Prednisone — Induction Chemotherapy: 100mg, oral administration on day 1 to 5 of each 3-week cycle until disease progression/stable disease after 2 cycles treatment, partial response after 4 cycles treatment or unacceptable toxicity develops, up to 6 cycles.
  Other Names: Prednisone Oral Product
Drug: Methotrexate — Induction Chemotherapy: 1g/m2, Intravenous administration on day 3 of each 3-week cycle from 2 to 5 cycles for patients with high recurrence risk of the central nervous system.
  Other Names: Methotrexate Injectable Solution

SUMMARY:
This is a prospective single-arm, multi-center, phase II clinical trial to observe the efficacy and safety of R-CHOP (Rituximab-Cyclophosphamide, Epirubicin, Vincristine and Prednisone) combined with lenalidomide in the first-line treatment for patients with medium to high risk/high risk diffuse large B cell lymphoma.

DETAILED DESCRIPTION:
Diffuse large B cell lymphoma (DLBCL) is the most common type of non-Hodgkin's lymphoma (NHL). Currently, R-CHOP is world-widely used in the first-line treatment for DLBCL. There are about one second of patients suffering relapse and drug resistance. Lenalidomide is an analog of thalidomide, the mechanism of anti-tumor action has not been fully elucidated. Lenalidomide has been proved to inhibit the proliferation of tumor cells in certain hematopoietic systems. At present, it has been approved for the treatment of multiple myeloma with good efficacy and safety. The goal of our trial is to assess the efficacy and safety of R-CHOP combined with lenalidomide in the first-line treatment for patients with medium to high risk/high risk diffuse large B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 70 years old (including 18 and 70)
2. Diagnosed as diffuse large B cell lymphoma
3. Subjects must be untreated (medium to high risk/high risk: International Prognostic Index (IPI) score 3-5 or aaIPI score 2-3/ Immunohistochemical staining of double expression (BCL2 ≥ 50% and C-MYC ≥ 40%) or P53 protein mutation positive ≥ 50%)
4. No receiving chemotherapy before enrollment
5. Having at least one measurable lesions
6. World health organization-Eastern Cooperative Oncology Group Performance Status (ECOG) 0-2
7. Life expectancy no less than 3 months
8. enough main organ function
9. Pregnancy test within 7 days must be negative for women of childbearing period, and appropriate measures should be taken for contraception for women in childbearing period during the study and six months after this study
10. Agreeing to sign the written informed consents

Exclusion Criteria:

1. Diagnosed as high-grade B-cell lymphoma, including non-specified and double-strike or triple-strike
2. Diagnosed as grey-zone lymphoma
3. Diagnosed as central nervous system lymphoma
4. Diagnosed as primary mediastinal large B-cell lymphoma
5. Diagnosed as CD20 negative diffuse large B-cell lymphoma
6. Other malignant tumor history or active malignant tumor need be treated
7. Serious surgery and trauma less than two weeks
8. Systemic therapy for serious acute/chronic infection
9. Congestive heart failure, uncontrolled coronary heart disease, arrhythmia and heart infarction less than 6 months
10. Vaccination with live attenuated vaccine less than 4 weeks
11. HIV-positive, AIDS patients and untreated active hepatitis
12. Patients with a history of deep vein thrombosis or pulmonary embolism less than 12 months
13. Patients with a history of mental illness
14. Researchers determine unsuited to participate in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-01-05 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-04-19 (Actual)

PRIMARY OUTCOMES:
2-year progression-free survival | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment
  the total proportion of patients with no progression from date of the first day of treatment to the date of confirmed progressive disease or death which one occurs first

SECONDARY OUTCOMES:
complete response rate | every 6 weeks from the day of the first cycle of induction chemotherapy treatment, up to 6 months after last patient's enrollment
  the total proportion of patients with complete response (CR)
2-year overall survival | from date of the first cycle of treatment to the date of death from any cause, assessed up to 2 years
  from date of first day of treatment to the date of death by any cause
incidence and relationship with study drugs of grade 3-4 adverse events | from the date of the first cycle of treatment to 6 months after last patient's enrollment
  the incidence and relationship with study drugs of grade 3 or 4 adverse events (based on NCI CTC-AE v4.03)

OTHER OUTCOMES:
exploratory endpoint | from the day of the first cycle of treatment to the date of confirmed progressive disease or death, whichever occurs first, up to 2 years after last patient's enrollment
  The correlation between hotspot driven gene mutations and complete response rate, PFS, or OS

CONTACTS AND LOCATIONS:
Overall Officials: Yanyan Liu, M.D. Ph.D, Study Director — Henan Cancer Hospital
Locations (1):
- Henan Cancer Hospital/The affiliated Cancer Hospital of ZhengZhou university, Zhengzhou, Henan, China